CLINICAL TRIAL: NCT07208370
Title: Outcome Predictors of Gillian Barrie Syndrome In Pediatrics
Brief Title: Outcomes of Gillian Barrie Syn
Acronym: mEGOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nourhan Maher Fawzy, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Outcomes of Gillian barrie Syn
Record Dates: First submitted 2025-09-15; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Outcome of Gillian Barrie

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GBS Group (Experimental)
  Interventions: Other: clinical assessment

INTERVENTIONS:
Other: clinical assessment — standraized clinical evaluation to assess disease sevirity and progration

SUMMARY:
This study analyze clinical and biological factors influencing disease course and outcome. Some research identified factors like disease severity, sensory symptoms, and autonomic instability as indicators of poor outcome. Ongoing research aims to develop accurate predictive models for improved treatment and care.

DETAILED DESCRIPTION:
Guillain-Barré Syndrome (GBS) is the most common cause of acute flaccid paralysis in children worldwide, often presenting with progressive weakness, areflexia, and varying degrees of autonomic and cranial nerve involvement. It is an immune-mediated disorder, commonly triggered by preceding infections such as Campylobacter jejuni, cytomegalovirus, or Epstein-Barr virus. Pediatric patients generally have a better prognosis than adults, yet a significant proportion still suffer from residual weakness or prolonged recovery. Understanding early predictors of outcome is essential for optimizing treatment and counseling families.[1][2] Several clinical and laboratory factors have been identified as potential predictors of poor outcomes in pediatric GBS. These include rapid progression to peak weakness, requirement of mechanical ventilation, presence of cranial nerve involvement (especially bulbar palsy), autonomic dysfunction, and the axonal subtypes of GBS on nerve conduction studies. Early identification of such factors allows for more aggressive supportive care and closer monitoring.[3][4][5] Electrophysiological classification also plays a vital role in predicting outcomes. Children with acute motor axonal neuropathy (AMAN) and acute motor-sensory axonal neuropathy (AMSAN) tend to have a slower and less complete recovery compared to those with acute inflammatory demyelinating polyneuropathy (AIDP). Furthermore, delayed initiation of immunotherapy such as intravenous immunoglobulin (IVIG) or plasma exchange may be associated with poorer prognosis.[6][7] Biomarkers like elevated cerebrospinal fluid (CSF) protein without pleocytosis (albuminocytologic dissociation) are typical in GBS but do not necessarily predict outcome. However, higher CSF protein levels in the early phase may correlate with more severe disease. Some recent studies have also suggested that MRI enhancement of spinal nerve roots may be associated with disease severity, although its prognostic value remains under investigation.[8][9] In conclusion, recognizing early outcome predictors in pediatric GBS is crucial for timely intervention, resource allocation, and family support. Although many children recover fully, identifying those at risk for complications can improve both short- and long-term care strategies.[2][3][10]

ELIGIBILITY:
Inclusion Criteria:

* All Pediatric patients (1 month to 18 years old) admitted with acute flaccid ascending paralysis and diagnosed as GBS.

Consent obtained from parents or legal guardians for participation and follow-up.

Exclusion Criteria:

* Children with pre-existing neuromuscular disorders. Patients with incomplete medical records or those lost to follow-up. Cases diagnosed as chronic inflammatory demyelinating polyneuropathy (CIDP).

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Pediatric Patients with Guillain-Barré Syndrome Achieving Full Recovery within 3 Months | first 3 months after diagnosis
  Proportion of pediatric patients with Guillain-Barré Syndrome achieving full recovery, as assessed by the Hughes Functional Grading Scale, within 3 months of diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kalita J, Kumar M, Misra UK. Prospective comparison of acute motor axonal neuropathy and acute inflammatory demyelinating polyradiculoneuropathy in 140 children with Guillain-Barre syndrome in India. Muscle Nerve. 2018 May;57(5):761-765. doi: 10.1002/mus.25992. Epub 2017 Nov 7. PMID 29053890
- [Background] Koul RL, Alfutaisi A. Prospective study of children with Guillain-Barre syndrome. Indian J Pediatr. 2008 Aug;75(8):787-90. doi: 10.1007/s12098-008-0099-1. Epub 2008 Jun 25. PMID 18581067
- [Background] Rajabally YA, Uncini A. Outcome and its predictors in Guillain-Barre syndrome. J Neurol Neurosurg Psychiatry. 2012 Jul;83(7):711-8. doi: 10.1136/jnnp-2011-301882. Epub 2012 May 7. PMID 22566597
- [Background] Korinthenberg R. Acute polyradiculoneuritis: Guillain-Barre syndrome. Handb Clin Neurol. 2013;112:1157-62. doi: 10.1016/B978-0-444-52910-7.00036-2. PMID 23622324
- [Background] Shahrizaila N, Yuki N. Antiganglioside antibodies in Guillain-Barre syndrome and its related conditions. Expert Rev Neurother. 2011 Sep;11(9):1305-13. doi: 10.1586/ern.11.114. PMID 21864076